CLINICAL TRIAL: NCT05505188
Title: Predictive and Impact of Pain at 6 Months in Patients Treated With Radiotherapy for Head and Neck Cancer
Brief Title: Predictive and Impact of Pain After 6 Months of Radiotherapy, in Head and Neck Cancer
Acronym: DIP-CAOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-A01894-35
Record Dates: First submitted 2022-03-14; First posted 2022-08-17 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Neuropathic Pain; Anxiety Disorder/Anxiety State; Pain, Chronic; Alcohol Use Disorder; Psychoactive Substance Use; Sleep; Symptoms and Signs; Addiction Nicotine
Keywords: Head and neck cancer; pain; Quality of life; Addiction; Depression
MeSH Terms: conditions — Neuralgia; Anxiety Disorders; Chronic Pain; Alcoholism; Signs and Symptoms; Tobacco Use Disorder; Head and Neck Neoplasms; Pain; Behavior, Addictive; Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: The main objective is to calculate the percentage of patients with neuropathic pain 6 months after the end of the treatments and to analyze the link between this pain and addictions, asthenia, depression, and in a more global way on the quality of life of patients. This evaluation will be done using validated questionnaires and self-questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Population (Other): no arm, single cohort follow-up
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Self-questionnaires are completed by the patient at the time of this consultation:
  * Neuropathic pain: NPSI in screening
  * Anxiety/depression: HADS in screening
  * Quality of life: EORTC (QLQC30 and H&N43)
  * Fatigue: MFI-20 hese self-questionnaires will be retrieved by the Clinical Research Associate (CRA) for verification.
  Depending on the result of the NPSI questionnaire can be completed to better characterize neuropathic pain.
  Depending on the result of the HADS, the MADRS questionnaire can be completed to quantify the degree of depression.
  Individuals diagnosed with neuropathic pain or other depressive symptoms during the 6-month inclusion period will be referred to and managed by specialized practitioners. This assistance will be indicated in follow-up report

SUMMARY:
Head and neck cancers are a source of complications and after-effects related to the disease and treatment. These cancers and their treatment alter the quality of life of patients and generate pain with physical and psychological components. Chronic pain affects 36% of patients at 6 months and 30% after this period. These pains are responsible for the consumption of level II and III analgesics in 53% of these patients. At the same time, after the end of treatment, nearly a quarter of patients continued to smoke and half still consumed alcohol at least twice a week.

The hypothesis of this research is to investigate the correlation between pain and the continuation of addictions, the occurrence of depressive states, asthenia and the alteration of the patients' global quality of life.

The investigators propose a two-center prospective cohort study to evaluate this hypothesis at 6 months after radiotherapy treatment.

This study is planned to include 120 patients with a first head and neck cancer whit radiotherapy as part of their treatment sequence. The expected duration of inclusion is 18 months.

The identification of factors affecting survival, quality of life and patient compliance is essential to determine appropriate management, particularly by creating appropriate therapeutic education programs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a first Head and neck cancer whose therapeutic sequence involves radiotherapy
* Patient over 18 years of age
* Having given written consent
* patient not previously treated with radiotherapy
* Life expectancy > 3 months
* World Health Organization (WHO) score < 3
* Histologically proven Head and Neck cancer
* Stable patient, with no signs of recurrence or other progressive neoplasia at the time of the examination
* Patient treated with radiotherapy
* Patient fluent in French

Exclusion Criteria:

* Non-consenting patient
* History of malignancy, other than treated and cured basal cell or cervical cancer
* Patient who has had a salvage surgery other than lymph node removal
* Patient with evidence of recurrence or other progressive neoplasia at the time of examination
* Patient who has had previous mutilating surgery (causing sequelae of swallowing and eating)
* Uncontrolled infectious pathology
* Patient under 18 years of age
* Patient who is not fluent in French
* Patient with a psychiatric pathology that could disrupt the study or prevent the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
change, neuropathic pain 1 | Day 0", "Month 6"
  Neuropathic Pain Symptom Inventory (NPSI) questionnaire, score 0 to 10, higher scores mean a worse, score 0 to 100, higher scores mean a worse outcome

SECONDARY OUTCOMES:
change, anxiety/depression | Day 0", "Month 6"
  with Hospital Anxiety and Depression Scale (HADS), score 0 to 21, higher scores mean a worse outcome
change, anxiety/depression 1 | Day 0", "Month 6"
  Montgomery and Asberg Depression Scale (MADRS) questionnaire, score 0 to 60, higher scores mean a worse outcome
change, quality of life | Day 0", "Month 6"
  QLQC30 questionnaire of Quality of Life, score 30-100, higher scores indicating better outcomes. the questionnaire measures several factors: physical fitness, professional activity, pain, nutrition, secondary effect, psychological and social status.
change, quality of life 1 | Day 0", "Month 6"
  H&N43 questionnaire of Quality of Life, score 43 to 172, higher scores indicating a worse outcomes. The questionnaire measures several factors:secondary effect, self-image, sociability, sexuality.
change, fatigue | Day 0", "Month 6"
  Multidimensional Fatigue Inventory (MFI-20) questionnaire, score 20 to 100, high scores represent more fatigue
change, symptoms related to head and neck cancer | Day 0", "Month 6"
  MD Anderson Symptom Inventory Head and Neck (MDASI-HN) questionnaire, score 0 to 220, higher scores indicating more symptoms
change, sleep | Day 0", "Month 6"
  question about sleep quality 0-10, higher scores indicating better outcomes
change, the impact of pain | Day 0", "Month 6"
  short pain questionnaire in French (QCD), score 0 to 120, high scores represent more impact of pain
change, Alcohol Use and Consumption Disorder | Day 0", "Month 6"
  Diagnostic and statistical manual of mental disorders (5th ed.) (DSM5) , questionnaire, score 0 to 115, high scores represent more disorder
change use of other psychoactive substances | Day 0", "Month 6"
  Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) alcool questionnaire, score 0 to 39, high scores represent more addiction
change severity of nicotine addiction | Day 0", "Month 6"
  Fagerström questionnaire, score 0 to 10, high scores represent more addiction

CONTACTS AND LOCATIONS:
Overall Officials: maxime humbert, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No